CLINICAL TRIAL: NCT06814795
Title: Feasibility of Medically Tailored Meals for Pediatric Populations at Risk for Disparities in Serious Illness Outcomes Due to Inequities in Social Drivers of Health (MTM-Kids)
Brief Title: Medically Tailored Meals for Kids
Acronym: MTM-Kids
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: LCCC2427; R21NR021288 (NIH)
Record Dates: First submitted 2025-01-17; First posted 2025-02-07 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Pediatric Cancer
Keywords: chemotherapy-induced alterations in taste; Food insecurity; Nutrition insecurity; Household material hardship; Resource hardship; Social drivers of health disparities
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Feasibility of study processes and the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Medically-tailored meals for children being treated for cancer with chemotherapy (Experimental): The intervention will be 12-weeks induration, with weekly "doses" (meal deliveries) of up to 10 healthy, frozen meals per week for household use as needed, plus selected condiments for personalization.
  Interventions: Other: Medically tailored meals

INTERVENTIONS:
Other: Medically tailored meals — The intervention will be 12-weeks in duration, with "doses" (meal deliveries) of up to 10 healthy, frozen meals per week for household use as needed, plus selected condiments for personalization
  Other Names: MTM-Kids

SUMMARY:
The purpose of this project is to learn whether an intervention that provides households with home-delivered healthy, frozen meals tailored to illness related conditions for 12 weeks during a child's treatment for serious illness is feasible and acceptable to the child and parent mainly responsible for the child's care.

DETAILED DESCRIPTION:
Food insecurity (uncertainty about having enough food for the household) and nutrition insecurity (uncertainty about access and affordability of foods that promotes health and quality of life [QOL]) are clinically-relevant, actionable social drivers of health (SDOH) disparities for pediatric (age 0-17.9 years) populations. Food and nutrition insecurity are especially relevant in pediatric populations vulnerable to disparities in outcomes of serious illnesses (life-threatening illnesses with taxing symptoms, treatments, and caregiving requirements). Pediatric cancer is an example. Children living in poverty with associated adverse SDOH are less likely survive either highly treatable cancers, or high-risk cancers that require regimens with costly targeted immunotherapy to optimize prospects for survival.. Poor nutrition increases risk of infection and poorer treatment tolerance, QOL, daily functioning and treatment responsiveness. Food-related insecurities may partly account for links between household poverty and poorer outcomes, and for the accelerated biological aging observed in pediatric and young adult cancer survivors. Moreover, poor eating habits developed treatment can persist into survivorship to heighten risks for secondary cardio-vascular conditions and cancers. Research on serious illness-related cost-coping suggests that parents and other primary caregivers legally and financially responsible for meeting the child's medical and day-to-day needs (hereafter "parents") may stretch food dollars by purchasing low priced, processed food with poor nutritional value. These purchasing choices contribute to household nutrition insecurity. Processed foods are also easy to prepare and thus appeal to parents who juggle time demands of complex caregiving and usual social roles. Because of chemotherapy-induced alterations in taste, these foods also appeal to young patients who crave food high in sugar and/or sodium. Parents and siblings may go without food and other essentials (needed health or dental care, prescribed medications [insulin], health insurance) to conserve the household's monetary assets to meet the needs of the child who is ill; these decisions heighten parent and sibling vulnerabilities to poorer health and QOL. In pediatric cancer, one approach being studied to address outcome disparities driven by food-related insecurities is to provide the household with gift cards for an online grocery delivery platform. Card amount is determined by household size and minimal cost for the Thrifty Food Plan per United States Department of Agriculture (USDA). No nutritional guidance is provided and parental time demands may limit their capacity to prepare healthy meals. To address health disparities in households experiencing food-related insecurities in the context of serious pediatric illness, holistic models that embed equity in care delivery by integrating food and nutrition interventions with state-of-the-science clinical care to address adverse SDOH are needed. Medically tailor meals (MTM) offer a Food is Medicine approach to addressing health disparities in pediatric serious illness populations. MTM comprise home-delivered meals tailored to medical needs of individuals with at risk for health disparities and barriers to preparing healthy food. In studies of adults, MTM interventions were associated with better health outcomes and less health care spending. Here, the investigators propose Medically-Tailored Meals for Kids (MTM-Kids), an extension of the MTM concept to pediatric serious illness populations for whom SDOH inequities affect outcomes, using pediatric cancer as the proof of concept. MTM-Kids account for nutritional needs, chemotherapy-induced alterations in taste, and illness-related financial burden and time demands. The purpose of the investigation is to determine feasibility of the MTM-methods and intervention for a future efficacy trial to improve food and nutrition security for children at risk for poorer outcomes due to SDOH inequities. The investigators will work with Equiti Foods, a small social enterprise that makes tasty, healthy, and culturally conscious frozen meals with start-up funding from National Institutes of Minority Health and Health Disparities. The primary research question is, "For households experiencing related insecurities, is providing healthy, frozen meals tailored to chemotherapy-induced alterations in taste feasible, appropriate and acceptable to children in active treatment for cancer and their parents?". After tailoring flavorings of the existing healthy, frozen means, the investigators will: 1. determine the feasibility, appropriateness, acceptability and accessibility of MTM-Kids; and 2. identify signals of change in food-related insecurities, cost coping, parental role demands and financial well-being. The investigation will be guided by the CONSORT extension for feasibility studies. Quantitative and qualitative feedback at multiple time points will enable rapid refinements of the MTM-Kids program and protocol for the future efficacy trial. The results will inform the potential for a future 2-group randomized efficacy trial with gift cards for an online grocery home delivery website as the likely comparator, and later cost effectiveness studies that advance our goal to extend healthcare financing models to include MTM in pediatric healthcare settings where seriously ill children receive care.

ELIGIBILITY:
Inclusion Criteria:

Eligible children (n=15) will:

* be under the care of The University of North Carolina at Chapel Hill School of Medicine, Department of Pediatrics, Division of Pediatric Hematology/Oncology
* have completed at least one cycle of cancer chemotherapy that included an agent known to cause alterations in taste,
* expect to undergo at least two more cycles,
* be aged 12-17.9 years
* communicate in English or Spanish.

Eligible adults (n=15) will:

* be the primary parental caregiver of a study-eligible child,
* be aged 18 years or older
* communicate in English or Spanish.

Exclusion Criteria:

* none if inclusion criteria are met

Ages: 12 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Parent-reported feasibility, acceptability, appropriateness and accessibility of MTM-Kids | Baseline and 12 weeks
  Each domain will be measured by 4-items developed by others and adapted for this study. Parents will be asked to read each item and indicate their response using 5-point scales anchored by 1=completely disagree and 5=completely aDomain scores will be calculated by summing item responses and dividing the sum by 4. Domain score range is 1-higher scores indicating better MTM program feasibility, acceptability, appropriateness and accessibility.
Adolescent-reported acceptability and appropriateness of MTM-Kids | Baseline and 12 weeks
  Each of these two domains of feasibility will be measured using items developed and validated by others and adapted for this study. Each domain has 4-items. Adolescents will be asked to read each item and indicate their response using scales anchored by 1=completely disagree and 5=completely agree. Domain scores will be calculated by summing responses and dividing the sum by 4. Domain score range is 1-4, with higher scores indicating better acceptability appropriateness

OTHER OUTCOMES:
Parent-reported household food insecurity | Baseline and 12 weeks
  Measured by the 6-item Food Security Scale. Parents will be asked to indicate whether they experienced the condition during the past 3 month and, in some cases, how often. Scores will be estimated by counting the number of affirmative responses (yes, sometimes, or often); these scores can be categorized, such that 0-1=very low food insecurity, 2-4food insecurity, and 5-6=high food insecurity.
Parent-reported household nutrition insecurity | Baseline and 12 weeks
  Measured by the 4-item Nutrition Security Scale plus 2 items from the Healthfulness Choice Scale. Parents will be use a 5-point scale, anchored by 1=never and 5=always, plus a don't know/prefer not to answer option. Scores will estimated by counting the number of affirmative responses (sometimes, often, or always); these scores can be categorized such that 0-1=very low nutrition insecurity, 2-4= low nutrition insecurity, and 5-6=high nutrition insecurity
Parental role demands | Baseline and 12 weeks
  Measured with a set of Patient-Reported Outcome Measurement System v.2 (PROMIS v.2) items that ask about satisfaction with perceived social role performance. Parents will be asked to respond to the PROMIS items using a scale anchored by 1=not at all and 5=very much. Item responses will be summed and scored using the T-score metHigher scores indicate greater satisfaction with social role performance.
Parental financial coping behaviors | Baseline and 12 weeks
  Measured by 7 questions from the Financial Coping Behaviors Scale currently being asked in a study of financial distress during treatment of pediatric acute lymphoblastic leukemia (ALL; ACCL20N1CD). Parents participating in MTM-Kidonly be asked about financial coping strategies with implications for the health of the adolescent or another family member. Parents will be asked to use a 3-point response scale anchored by 0=never and 2=several times) to indicate how often they used each coping behavior in the prior month. Item responses will be summed for a total score that can range from 0-14. (higher scores indicate use of more types of financial coping behaviors)
Parental financial well-being | Baseline and 12 weeks
  Measured by the 8-item Personal Financial Well-being Scale (PFWS).The PFWS uses a 10-point response scale. Scores are calculated by summing item responses and dividing by 8. Scores can range from 1 to 10, with 1 indicating poorest wellbeing and 10 indicating highest financial wellbeing. The PFWS has undergone rigorous psychometric testing to establish validity of the latent construct, psychometric properties and norms.
Adolescent chemotherapy-induced alterations in taste | Baseline and up to 12 weeks
  Measured by 13-items from the Chemotherapy-Induced Alterations in Taste Scale (CiTAS). Adolescents will be ask to use a 5-point scale to indicate how much the taste change bothered them this week. Scores will be calculated by summing item responses and dividing by 13 (lower scores indicate less alteration in taste).
Adolescent-reported other chemotherapy-related symptoms | Baseline and up to 12 weeks
  Measured by the 15-item Symptom Screening in Pediatrics (SSPedi) tool. Adolescents will be asked to use a 5-point response scale anchored by 0 (not at all) and 4 (worst bother) to indicate how much each symptom bothered them today or yesterday Scores will be calculated by summing item responses. Scores can range from 0-60 (lower scores indicate less symptom severity)

CONTACTS AND LOCATIONS:
Overall Officials: Sheila J. Santacroce, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- North Carolina Basnight Cancer Hospital, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication of primary paper and for 5 years thereafter
Access Criteria: Local Institutional Review Board (IRB)-approved application for proposed secondary analyses

REFERENCES:
- [Background] Coleman-Jensen A, Rabbitt MP, Gregory CA, Singh A. Household Food Security in the United States inU.S. Department of Agriculture Economic Research Service. Washington, D. C. 2022.
- [Background] Mozaffarian D. Measuring and addressing nutritional secutiry to achieve health and health equity HeAffairs Health Policy Brief. March 30, 2023. https://doi.org/10.1377/hpb2023216.92558
- [Background] American Academy of Pediatrics Council on Community Pediatrics. Poverty and child health in the UStates. Pediatrics. 2016;137:e20160339. https://doi.org/10.1542/peds.2016-0339
- [Background] Zenk SN, Tabak LA, Perez-Stable EJ. Research Opportunities to Address Nutrition Insecurity and Disparities. JAMA. 2022 May 24;327(20):1953-1954. doi: 10.1001/jama.2022.7159. No abstract available. PMID 35486390
- [Background] Kelley AS. Defining "serious illness". J Palliat Med. 2014 Sep;17(9):985. doi: 10.1089/jpm.2014.0164. Epub 2014 Aug 12. No abstract available. PMID 25115302
- [Background] Bona K, Blonquist TM, Neuberg DS, Silverman LB, Wolfe J. Impact of Socioeconomic Status on Timing of Relapse and Overall Survival for Children Treated on Dana-Farber Cancer Institute ALL Consortium Protocols (2000-2010). Pediatr Blood Cancer. 2016 Jun;63(6):1012-8. doi: 10.1002/pbc.25928. Epub 2016 Feb 23. PMID 26913850
- [Background] Wadhwa A, Chen Y, Hageman L, Hoppmann A, Angiolillo A, Dickens DS, Neglia JP, Ravindranath Y, Ritchey AK, Termuhlen A, Wong FL, Landier W, Bhatia S. Poverty and relapse risk in children with acute lymphoblastic leukemia: a Children's Oncology Group study AALL03N1 report. Blood. 2023 Jul 20;142(3):221-229. doi: 10.1182/blood.2023019631. PMID 37070673
- [Background] Bona K, Li Y, Winestone LE, Getz KD, Huang YS, Fisher BT, Desai AV, Richardson T, Hall M, Naranjo A, Henderson TO, Aplenc R, Bagatell R. Poverty and Targeted Immunotherapy: Survival in Children's Oncology Group Clinical Trials for High-Risk Neuroblastoma. J Natl Cancer Inst. 2021 Mar 1;113(3):282-291. doi: 10.1093/jnci/djaa107. PMID 33227816
- [Background] Barr RD, Gomez-Almaguer D, Jaime-Perez JC, Ruiz-Arguelles GJ. Importance of Nutrition in the Treatment of Leukemia in Children and Adolescents. Arch Med Res. 2016 Nov;47(8):585-592. doi: 10.1016/j.arcmed.2016.11.013. PMID 28476186
- [Background] Tripodi SI, Bergami E, Panigari A, Caissutti V, Brovia C, De Cicco M, Cereda E, Caccialanza R, Zecca M. The role of nutrition in children with cancer. Tumori. 2023 Feb;109(1):19-27. doi: 10.1177/03008916221084740. Epub 2022 Jun 19. PMID 35722985
- [Background] Berkowitz SA, Palakshappa D, Seligman HK, Hanmer J. Changes in Food Insecurity and Changes in Patient-Reported Outcomes: a Nationally Representative Cohort Study. J Gen Intern Med. 2022 Nov;37(14):3638-3644. doi: 10.1007/s11606-021-07293-4. Epub 2022 Jan 6. PMID 34993877
- [Background] Pedretti L, Massa S, Leardini D, Muratore E, Rahman S, Pession A, Esposito S, Masetti R. Role of Nutrition in Pediatric Patients with Cancer. Nutrients. 2023 Jan 30;15(3):710. doi: 10.3390/nu15030710. PMID 36771416
- [Background] Orgel E, Framson C, Buxton R, Kim J, Li G, Tucci J, Freyer DR, Sun W, Oberley MJ, Dieli-Conwright C, Mittelman SD. Caloric and nutrient restriction to augment chemotherapy efficacy for acute lymphoblastic leukemia: the IDEAL trial. Blood Adv. 2021 Apr 13;5(7):1853-1861. doi: 10.1182/bloodadvances.2020004018. PMID 33792627
- [Background] Bhatia S, Landier W, Hageman L, Kim H, Chen Y, Crews KR, Evans WE, Bostrom B, Casillas J, Dickens DS, Maloney KW, Neglia JP, Ravindranath Y, Ritchey AK, Wong FL, Relling MV. 6MP adherence in a multiracial cohort of children with acute lymphoblastic leukemia: a Children's Oncology Group study. Blood. 2014 Oct 9;124(15):2345-53. doi: 10.1182/blood-2014-01-552166. Epub 2014 May 14. PMID 24829202
- [Background] Gomez-Almaguer D, Ruiz-Arguelles GJ, Ponce-de-Leon S. Nutritional status and socio-economic conditions as prognostic factors in the outcome of therapy in childhood acute lymphoblastic leukemia. Int J Cancer Suppl. 1998;11:52-5. doi: 10.1002/(sici)1097-0215(1998)78:11+3.0.co;2-3. PMID 9876479
- [Background] Wilder ME, Kulie P, Jensen C, Levett P, Blanchard J, Dominguez LW, Portela M, Srivastava A, Li Y, McCarthy ML. The Impact of Social Determinants of Health on Medication Adherence: a Systematic Review and Meta-analysis. J Gen Intern Med. 2021 May;36(5):1359-1370. doi: 10.1007/s11606-020-06447-0. Epub 2021 Jan 29. PMID 33515188
- [Background] Gehle SC, Kleissler D, Heiling H, Deal A, Xu Z, Ayer Miller VL, Taylor JA, Smitherman AB. Accelerated epigenetic aging and myopenia in young adult cancer survivors. Cancer Med. 2023 Jun;12(11):12149-12160. doi: 10.1002/cam4.5908. Epub 2023 Apr 9. PMID 37031460
- [Background] Smitherman AB, Wood WA, Mitin N, Ayer Miller VL, Deal AM, Davis IJ, Blatt J, Gold SH, Muss HB. Accelerated aging among childhood, adolescent, and young adult cancer survivors is evidenced by increased expression of p16INK4a and frailty. Cancer. 2020 Nov 15;126(22):4975-4983. doi: 10.1002/cncr.33112. Epub 2020 Aug 24. PMID 32830315
- [Background] Ogland-Hand C, Ciesielski TH, Daunov K, Bean MK, Nock NL. Food Insecurity and Nutritional Challenges in Adolescent and Young Adult Cancer Survivors in the U.S.A.: A Narrative Review and Call to Action. Nutrients. 2023 Apr 1;15(7):1731. doi: 10.3390/nu15071731. PMID 37049571
- [Background] McDougall JA, Jaffe SA, Guest DD, Sussman AL. The Balance Between Food and Medical Care: Experiences of Food Insecurity Among Cancer Survivors and Informal Caregivers. J Hunger Environ Nutr. 2022;17(3):380-396. doi: 10.1080/19320248.2021.1892295. Epub 2021 Feb 25. PMID 35757157
- [Background] Thom B, Benedict C, Friedman DN, Watson SE, Zeitler MS, Chino F. Economic distress, financial toxicity, and medical cost-coping in young adult cancer survivors during the COVID-19 pandemic: Findings from an online sample. Cancer. 2021 Dec 1;127(23):4481-4491. doi: 10.1002/cncr.33823. Epub 2021 Aug 5. PMID 34351638
- [Background] Nucci D, Santangelo OE, Provenzano S, Nardi M, Firenze A, Gianfredi V. Altered Food Behavior and Cancer: A Systematic Review of the Literature. Int J Environ Res Public Health. 2022 Aug 18;19(16):10299. doi: 10.3390/ijerph191610299. PMID 36011935
- [Background] Santacroce SJ, Tan KR, Killela MK. A systematic scoping review of the recent literature ( approximately 2011-2017) about the costs of illness to parents of children diagnosed with cancer. Eur J Oncol Nurs. 2018 Aug;35:22-32. doi: 10.1016/j.ejon.2018.04.004. Epub 2018 May 17. PMID 30057080
- [Background] Downer S, Clippinger E, Kummer C. Food is Medicine research action plan. Published Jan. 27, 2022.
- [Background] Hager K, Cudhea FP, Wong JB, Berkowitz SA, Downer S, Lauren BN, Mozaffarian D. Association of National Expansion of Insurance Coverage of Medically Tailored Meals With Estimated Hospitalizations and Health Care Expenditures in the US. JAMA Netw Open. 2022 Oct 3;5(10):e2236898. doi: 10.1001/jamanetworkopen.2022.36898. PMID 36251292
- [Background] Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA; PAFS consensus group. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. Pilot Feasibility Stud. 2016 Oct 21;2:64. doi: 10.1186/s40814-016-0105-8. eCollection 2016. PMID 27965879
- [Background] U.S. Department of Agriculture Economic Research Service. U.S. Household food security survey mothree-stage design, with screeners. 2012. https://www.ers.usda.gov/topics/food-nutrition-assistabcesecurity-in-the-u-s-/measurement
- [Background] Calloway EE, Carpenter LR, Gargano T, Sharp JL, Yaroch AL. Development of new measures to assess household nutrition security, and choice in dietary characteristics. Appetite. 2022 Dec 1;179:106288. doi: 10.1016/j.appet.2022.106288. Epub 2022 Aug 29. PMID 36049571
- [Background] Hahn EA, DeWalt DA, Bode RK, Garcia SF, DeVellis RF, Correia H, Cella D; PROMIS Cooperative Group. New English and Spanish social health measures will facilitate evaluating health determinants. Health Psychol. 2014 May;33(5):490-9. doi: 10.1037/hea0000055. Epub 2014 Jan 20. PMID 24447188
- [Background] Beauchemin M, Santacroce SJ, Bona K, Dang H, Alexander S, Allen K, De Los Santos C, Fisher B, Muneton-Castano Y, Ponce O, Vargas S, Sugalski A, Sung L, Parsons S. Rationale and design of Children's Oncology Group (COG) study ACCL20N1CD: financial distress during treatment of acute lymphoblastic leukemia in the United States. BMC Health Serv Res. 2022 Jun 28;22(1):832. doi: 10.1186/s12913-022-08201-0. PMID 35764995
- [Background] Prawitz A, et al.. InCharge Financial Distress/Financial Well-Being Scale: development, administrationscore interpretation. Financial Counseling & Planning. 2006;17 34-50 doi: doi:10.1037/t60365-000
- [Background] Dupuis LL, Johnston DL, Baggott C, Hyslop S, Tomlinson D, Gibson P, Orsey A, Dix D, Price V, Vanan M, Portwine C, Kuczynski S, Spiegler B, Tomlinson GA, Sung L. Validation of the Symptom Screening in Pediatrics Tool in Children Receiving Cancer Treatments. J Natl Cancer Inst. 2018 Jun 1;110(6):661-668. doi: 10.1093/jnci/djx250. PMID 29272441
- [Background] Kano T, Kanda K. Development and validation of a chemotherapy-induced taste alteration scale. Oncol Nurs Forum. 2013 Mar;40(2):E79-85. doi: 10.1188/13.ONF.E79-E85. PMID 23448748
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Derived] Thom B, Crowder VR, Smitherman AB, Cosgrove BS, Bosch R, Vardhan Y, Matt CN, Ammerman A, Santacroce SJ. Study protocol: Feasibility of medically tailored meals for pediatric populations at risk for disparities in serious illness outcomes due to inequities in food-related social drivers of health (MTM-Kids). PLoS One. 2025 Jul 31;20(7):e0326762. doi: 10.1371/journal.pone.0326762. eCollection 2025. PMID 40743050